CLINICAL TRIAL: NCT01731249
Title: A Randomised, Double-blind, Placebo-controlled, Multi-national, Phase IIIb Study to Assess the Sustained Clinical Effect and Safety of Sublingual Immunotherapy Administered as Birch Pollen Extract Solution at a Dose of 300 IR Once Daily to Patients Suffering From Birch Pollen-induced Rhinoconjunctivitis
Brief Title: Efficacy and Safety Study of a Sublingual Immunotherapy Solution to Treat Patients Suffering From Birch Pollen Allergic Rhinoconjunctivitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stallergenes Greer (Industry)
Collaborators: Quintiles, Inc. (Industry); Aptuit (Industry); Cenduit LLC (Industry); PHT Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VO68.10; 2010-020693-42 (EudraCT Number)
Record Dates: First submitted 2012-11-15; First posted 2012-11-21 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Hypersensitivity; Allergic Rhinitis; Allergic Conjunctivitis; Seasonal Allergy
Keywords: Sublingual immunotherapy; Birch pollen extract solution; Allergic rhinoconjunctivitis
MeSH Terms: conditions — Hypersensitivity; Rhinitis, Allergic; Conjunctivitis, Allergic; Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo sublingual solution
  Interventions: Biological: Placebo
- Birch pollen allergen extract (Experimental): Sublingual Solution of Birch pollen allergen extract 300IR once daily 5 months per year and during 2 years
  Interventions: Biological: Birch pollen allergen extract

INTERVENTIONS:
Biological: Placebo — 10 actuations of placebo sublingual solution once daily 5 months a year and during 2 years
  Arms: Placebo
Biological: Birch pollen allergen extract — Sublingual solution of Birch pollen allergen extract 300IR (10 actuations) once daily 5 months per year and during 2 years
  Other Names: Staloral Birch
  Arms: Birch pollen allergen extract

SUMMARY:
The purpose of this 2-year study is to assess the sustained clinical efficacy and safety of 300 IR/day of a sublingual solution of birch pollen allergen extract starting 4 months prior to the birch pollen season and continuing over the birch pollen season compared with placebo for reduction of rhinoconjunctivitis-related symptoms and anti-allergy medication usage.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic birch pollen-related allergic rhinoconjunctivitis for at least the previous 2 pollen seasons requiring intake of symptomatic treatment.
* Sensitization to birch pollen demonstrated by a positive Skin Prick Test to birch pollen with wheal diameter > 3 mm and birch pollen allergens specific IgE levels ≥ 0.70 kU/L.
* RRTSS based on the previous or on the penultimate birch pollen season ≥ 12 out of a maximum possible score of 18.
* Patients with an FEV1 (Forced Expiratory Volume at one second) ≥ 80% of the predicted value.
* Patients who are willing to comply with the protocol.
* Patients having given a signed informed consent before completing any study related procedure.

Exclusion Criteria:

* Patients with symptoms of rhinitis/rhinoconjunctivitis during the birch pollen season due to any other allergens (except alder and hazel). This includes patients with symptomatic allergic rhinitis/rhinoconjunctivitis due to cat or dog allergens, and living with these animals at home or at risk of frequent contacts with these animals (family, friends etc.) during the course of the study.
* Patient who previously received desensitization treatment to birch pollen and/or another Betulaceae sp. (for example hazel or alder) within the previous 5 years.
* Patients with ongoing treatment by immunotherapy with another allergen.
* Pregnancy (positive pregnancy test), breast-feeding.
* Female patients of childbearing potential planning a pregnancy during this study or not using a medically accepted contraceptive method (hormonal birth control [orally, injectable or by implant, for at least 2 months before enrolment], intrauterine device, spermicide used with a male condom, bilateral tubal ligation, diaphragm with spermicide, female condom, monogamous relationship with a vasectomised partner).
* Patients planning to move during the study or planning to leave the area during the birch pollen season for more than 1 week (7 consecutive days).
* Patients with moderate or severe persistent asthma (GINA 3 or 4).
* Patients with seasonal mild persistent asthma (GINA 2) necessitating treatment with inhaled glucocorticosteroids at a dose level greater than 400 mcg budesonide dose-equivalents.
* Patients with any nasal or oral condition that could interfere with the efficacy or safety assessments (such as nasal polyposis or oral inflammation).
* Patients with severe immune deficiency.
* Patients with a past or current disease, which as judged by the Investigator, may affect the patient's participation in or outcome of this study.
* Any other disease or condition which would place a patient at undue risk by being included in the study (according to the Investigator's opinion).
* Usual contra-indications of immunotherapy such as concomitant beta-blocker therapy whatever the route and/or immunosuppressive drugs.
* Patients treated with inhaled/systemic steroids (whatever the indication) within 4 weeks prior to Visit 1 (Screening), or with long acting systemic corticosteroids 12 weeks before Visit 1 (Screening).
* Patients under continuous corticotherapy (inhaled or systemic drugs).
* Patients following a strict low sodium diet as the study treatment contains 590 mg of sodium chloride per vial in a 10 mL solution.
* Investigators, co-Investigators, as well as their children or spouses and all study collaborators.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 574 (Actual)
Dates: Start 2010-11; Primary Completion 2012-07 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Average Adjusted Symptom Score | Year 2 of treatment
  Symptom score adjusted on patient's rescue medication usage

SECONDARY OUTCOMES:
Average Rhinoconjunctivitis Total Symptom Score | Year 2 of treatment
Average Rescue Medication Score | Year 2 of treatment
Each of Six Individual Average Rhinoconjunctivitis Symptom Scores | Year 2 of treatment
Average Combined Score | Year 2 of treatment
Average Rhinoconjunctivitis Visual Analogue Scale Score | Year 2 of treatment
Average Adjusted Visual Analogue Scale Score | Year 2 of treatment
Rescue Medication Usage | Year 2 of treatment
Proportion of Symptom-controlled Days | Year 2 of treatment
Rhinoconjunctivitis Quality of Life Questionnaire | Year 2 of treatment
Global evaluation of the efficacy by the patient | Year 2 of treatment
Sensitization profile | Before and after each treatment period (over 2 years)
  sensitization profile (mono- vs poly-sensitized) is derived from the skin prick test results
Asthma | Before, during and after each pollen season (over 2 years)
Immunological markers specific for birch pollen | Before and after each treatment period (over 2 years)
Economical Evaluation | Year 2 of treatment
  Proportion of days-off due to birch pollen-induced symptoms
Wheal diameter of the birch allergen Skin prick test | Before and after each treatment period (over 2 years)
Oral Provocation Test | Year 2 of treatment
  Analysis on a subset of patients presenting an Oral Allergy Syndrome at study entry
Mucosa Local Inflammation | Year 1 of treatment
  Analysis on a subset of patients
Safety assessments | ~20 months
  adverse events, physical examination including vital signs and laboratory data described by number of patients in each treatment group
Average adjusted Symptom score analysis by tertiles | Year 2 of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Margitta WORM, MD, PR, Principal Investigator — Allergie-Centrum-Charité, Klinik für Dermatologie, Venerologie und Allergologie, Charité Campus Mitte, Universitätsmedizin, Charitéplatz 1, 10117 Berlin, Germany
Locations (11):
- Alergologicka ordinace, Pilsen, Czechia
- National University Hospital - Allergy Unit 4222, Copenhagen, Denmark
- Merekivi Perearstid OÜ, Tallinn, Estonia
- Helsingin yliopistollinen keskussairaala, Helsinki, Finland
- NHC, Hôpitaux Universitaires de Strasbourg, Strasbourg, France
- Universitätsmedizin Berlin - Allergie-Centrum-Charité, Berlin, Germany
- Centre of Investigations and Treatment of Allergic Diseases, Riga, Latvia
- Allergic Diseases Diagnostics and Treatment Centre, Vilnius, Lithuania
- SPZOZ Uniwersytecki Szpital Kliniczny Nr 1im.N.Barlickiego w Uniwersystetu Medycznego w Łodzi, Lodz, Poland
- Imunologicko-alergologicka amb., Banská Bystrica, Slovakia
- Sahlgrenska Universitetssjukhuset - Avd för Lungmedicin och Allergi, Gothenburg, Sweden

REFERENCES:
- [Derived] Worm M, Rak S, de Blay F, Malling HJ, Melac M, Cadic V, Zeldin RK. Sustained efficacy and safety of a 300IR daily dose of a sublingual solution of birch pollen allergen extract in adults with allergic rhinoconjunctivitis: results of a double-blind, placebo-controlled study. Clin Transl Allergy. 2014 Feb 11;4(1):7. doi: 10.1186/2045-7022-4-7. PMID 24517417